CLINICAL TRIAL: NCT02163239
Title: Post Market Study: Use of the Reusable FloShield 10mm Endoscopic Cannula and Blunt Obturator and the Robotic FloShield System During Robot-assisted Laparoscopic Single-Site Surgery. A Multicenter Historical Control Comparison
Brief Title: Post Market Study for FloShield 10mm Reusable Cannula and Blunt Obturator and Robotic FloShield
Status: Terminated | Type: Observational
Why Stopped: Not meeting primary objective of the study
Sponsor: Minimally Invasive Devices, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FRT-0001
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Cholecystectomy; Benign Hysterectomy; Salingo-oophorectomy
Keywords: FloShield; MID; Minimally invasive surgery; Minimally Invasive devices; Robot-assisted Laparoscopic Surgery; Single-site Laparoscopic Surgery; Single Incision Laparoscopic Surgery; Cannula; Blunt Obturator; Cholecystectomy; Benign hysterectomy; Salpingo-oophorectomy
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 10mm Cannula: Subjects that are scheduled for a robot-assisted laparoscopic single-incision surgery for cholecystectomy, benign hysterectomy or salpingo-oophorectomy under the care of the study investigator
  Interventions: Device: Cannula and Blunt Obturator

INTERVENTIONS:
Device: Cannula and Blunt Obturator — The FloShield 10mm Endoscopic Cannula and Blunt Obturator will be used to maintain access to the peritoneal cavity during robot-assisted single site laparoscopic surgery
  Other Names: FloShield 10mm Endoscopic Cannula, FRT10C; FloShield Blunt Oburator, FRT10B

SUMMARY:
This study evaluates the use of the FloShield System with the FloShield 10mm reusable Cannula and Oburator during standard robotic laparoscopic single-site surgery. The study will evaluate the compatibility of the FloShield 10mm Cannula and Oburator with the daVinci® Robotic Surgical System during single-site laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Scheduled for a laparoscopic single-incision surgery for cholecystectomy, benign hysterectomy or salpingo-oophorectomy under the care of the study investigator
* Suitable candidate for surgery
* Is able to read and understand the informed consent form and has voluntarily provided written informed consent

Exclusion Criteria:

* Unfit for surgery: concomitant disorders incompatible with the study or surgery (at the discretion of the investigator)
* Subjects with known allergy (hypersensitivity) to Docusate Sodium
* Use of Surgiquest AirSeal during the laparoscopic single-site surgery
* Use of humidified insufflation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from a population of patients who are from the medical practice of the study investigator and who are scheduled to undergo robot-assisted laparoscopic single-incision surgery for cholecystectomy, benign hysterectomy or salpingo-oophorectomy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Completion rate | 1 - 4hr (Initial insertion to final withdrawal of the laparoscope)
  Completion rate is the percentage of users who successfully complete the task without critical errors. A critical error is defined as an error that results in an incorrect or incomplete outcome (Grade 1 and 2). In other words, the completion rate represents the percentage of participants who, when they are finished with the specified task, have an "output" that is correct (Grade 3 - 5). Note: If a participant requires assistance in order to achieve a correct output then the task will be scored as a critical error and the overall completion rate for the task will be affected. A completion rate of 90% is the goal for each task in this usability test.

SECONDARY OUTCOMES:
Performance | 1 - 4hr (Initial insertion to final withdrawal of the laparoscope)
  The secondary outcome from the study will be an assessment of the performance of the FloShield 10mm Cannula and Oburator/FloShield System in its ability to defog and clean the laparoscopic lens.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Poll, MD, Study Director — Minimally Invasive Devices
Locations (1):
- Baptist Health South Florida, Miami, Florida, United States